CLINICAL TRIAL: NCT00218673
Title: Randomized Controlled Trial of Russian IDU Peer Network HIV Prevention Intervention
Brief Title: RCT of Russian IDU Peer Network HIV Prevention Intervention - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Carl Latkin, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DESPR DA016142; 5R01DA016142 (NIH); R01-16142-1; NIDA-16142-1
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: HIV Infections
Keywords: HIV; injection drug use; social networks
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- experimental (Experimental): social network
  Interventions: Behavioral: Peer mentor intervention
- control (No Intervention): testing and counseling

INTERVENTIONS:
Behavioral: Peer mentor intervention — groups sessions, 8
  Arms: experimental

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial to assess the efficacy of a peer-educator intervention focused on injection drug users and their drug and sexual networks. We expect that participants who receive the intervention will demonstrate a reduction in the rate of HIV infection and HIV risk behaviors and members of their risk network will also demonstrate reductions in risk behaviors compared to those in the control group.

DETAILED DESCRIPTION:
Intravenous drug use (IDU) is driving the HIV epidemic in Russia; over 90% of all HIV-1 infections have occurred within communities of IDUs. In St. Petersburg (population 5 million), the prevalence of HIV infection in IDUs (estimated population 100,000) leapt from 4% in 1999 to 12% in 2000. At present there are an estimated 5-7 million IDUs, a four-fold increase since the end of the Soviet Union. In St. Petersburg, there has been a three-fold increase in regular IDUs and a nine-fold increase in teenage IDUs during the past five years.

The intervention to be tested in this study draws upon theoretical and empirical evidence suggesting that peer educator programs can have significant effects on the risk-related behaviors of both the educators and the peers whom they educate. Providing peer educator training to IDUs may efficiently cultivate sustainable protective behavioral norms related to injection and sexual risk among the IDU educators' social networks. Prior studies have demonstrated that peer educator programs can realize such normative changes, and it is hypothesized in this study that these normative changes will be reflected in significant reductions in the rates of HIV transmission among the peer educators and the members of their social networks.

Comparison condition: Informed by the Centers for Disease Control model of best practice" standard of care of HIV testing and counseling, participants in the comparison condition will receive risk reduction education and motivational counseling to reduce their risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Of legal age to independently provide written informed consent for research
* Report having injected drugs at least 12 times in the last three months
* HIV seronegative (ELISA confirmed)
* Willing and able to recruit at least three HIV risk network members who are eligible for study participation

Exclusion Criteria:

* Prior or concurrent enrollment in the last 6 months in another HIV behavioral or biomedical prevention study
* Psychological disturbance or cognitive impairment that appears to limit the ability to understand study procedures, as determined by clinic staff
* Any other condition that, in the opinion of the investigator, would make participation in the study unsafe, or otherwise interfere with the study objectives

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2003-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Incident number of HIV Infections in social networks | 1 year

SECONDARY OUTCOMES:
Self reported risk behaviors: entry into drug treatment, cessation of drug use | 1 year
Self reported risk behaviors: number of sex partners, freq of condom use | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Carl Latkin, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Biomedical Center, Saint Petersburg, Russia

REFERENCES:
- [Derived] Hoffman IF, Latkin CA, Kukhareva PV, Malov SV, Batluk JV, Shaboltas AV, Skochilov RV, Sokolov NV, Verevochkin SV, Hudgens MG, Kozlov AP. A peer-educator network HIV prevention intervention among injection drug users: results of a randomized controlled trial in St. Petersburg, Russia. AIDS Behav. 2013 Sep;17(7):2510-20. doi: 10.1007/s10461-013-0563-4. PMID 23881187